CLINICAL TRIAL: NCT03867747
Title: Radiosurgery for the Treatment of Refractory Ventricular Extrasystoles and Tachycardias (RAVENTA)
Brief Title: Radiosurgery for the Treatment of Refractory Ventricular Extrasystoles and Tachycardias
Acronym: RAVENTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Collaborators: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Juergen Dunst, Prof., Prof. Dr. med. Juergen Dunst, University Hospital Schleswig-Holstein
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZKS-121-09
Record Dates: First submitted 2019-03-05; First posted 2019-03-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Ventricular Tachycardia
Keywords: Ventricular Tachycardia; Stereotactic Body Radiation Therapy; Radiosurgery
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cardiac Radiosurgery (Experimental): 25 Gy in a single fraction
  Interventions: Radiation: Cardiac Radiosurgery

INTERVENTIONS:
Radiation: Cardiac Radiosurgery — Image-guided stereotactic body radiation therapy

SUMMARY:
Patients with refractory ventricular extrasystoles or tachycardia not eligible for catheter ablation will receive single fraction stereotactic body radiation therapy (cardiac radiosurgery) with 25 Gy.

Investigators initiated this study to demonstrate that in at least 70% of the patients the planned cardiac radiosurgery may be performed without any interruption or treatment related interventional events within the first 30 days after treatment.

DETAILED DESCRIPTION:
Primary endpoint: 30-day post-intervention safety defined as presence of both, radiosurgery delivery of the planned dose to the intended target area, and no possibly treatment related serious adverse events in the first 30 days after treatment.

Secondary endpoints: evaluated at 1 year

* Changes in ventricular tachycardia episodes and ICD shocks
* Changes in antiarrhythmic medication due to treatment effects
* Occurrence of possibly treatment related adverse events in the first year after treatment
* Changes in patient-reported quality of life
* Overall survival
* Safety profile

ELIGIBILITY:
Inclusion Criteria:

* Patients with structural heart disease and implantable cardioverter defibrillator (ICD)
* Age > 18 years
* either

  1. Recurring symptomatic monomorphic ventricular tachycardia that requires ICD intervention (e.g. shock or anti-tachycardia stimulation). At least 3 episodes within the 3 months prior to inclusion or
  2. induction of symptomatic monomorphic ventricular tachycardia that requires ICD intervention (e.g. shock or anti-tachycardia stimulation). Induction triggered by ICD or during electrophysiology studies (EPS) or both, a) and b)
* Refractory to antiarrhythmic combination therapy
* Beside the cardiac conditions: No competing illness that would additionally limit the life expectancy to less than 6 months
* No prior radiation therapy in the thorax area
* No pregnancy and no active breastfeeding
* Ability to consent and consent to study participation

Exclusion Criteria:

* ICD electrode malfunction of ICD readings outside reference range
* Lack of evidence of a myocardial scar (Computer tomography or magnetic resonance tomography for MRI-capable ICD aggregates or electrophysiological measurement)
* No possible induction of symptomatic monomorphic ventricular tachycardia non-persistent or persistent with delivery of ICD therapies such as antitachycardic pacing or shock
* Contraindication to radiosurgery (e.g. precise target volume definition not possible due to image artifacts created from a left ventricular assist device (LVAD))
* Inability to consent or missing or withdrawn consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2024-10-20 (Actual)

PRIMARY OUTCOMES:
Acute toxicity analysed by Adverse Event (AE)- and Serious Adverse Event (SAE)-reports | 30 days after radiosurgery

SECONDARY OUTCOMES:
Late toxicity analysed by Adverse Event (AE)- and Serious Adverse Event (SAE)-reports | 12 months after radiosurgery
Ventricular tachycardia burden reduction analysed by number of episodes and ICD shocks | At the time of inclusion and 12 months after radiosurgery
Overall Survival | 12 months after radiosurgery
Quality of Life questionnaire | At the time of inclusion and 12 months after radiosurgery

CONTACTS AND LOCATIONS:
Overall Officials: Roland R Tilz, Prof., Principal Investigator — University Hospital Schleswig-Holstein; Juergen Dunst, Prof., Principal Investigator — University Hospital Schleswig-Holstein
Locations (6):
- Germany (6):
  - University Clinic Mannheim, Mannheim, Baden-Wurttemberg
  - Hospital of the Ludwig-Maximilians-University Munich, Munich, Bavaria
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - University Medical Center Schleswig-Holstein, Kiel, Schleswig-Holstein
  - University Medical Center Schleswig-Holstein, Lübeck, Schleswig-Holstein
  - University Medical Center Charite Berlin, Berlin

REFERENCES:
- [Background] Blanck O, Buergy D, Vens M, Eidinger L, Zaman A, Krug D, Rudic B, Boda-Heggemann J, Giordano FA, Boldt LH, Mehrhof F, Budach V, Schweikard A, Olbrich D, Konig IR, Siebert FA, Vonthein R, Dunst J, Bonnemeier H. Radiosurgery for ventricular tachycardia: preclinical and clinical evidence and study design for a German multi-center multi-platform feasibility trial (RAVENTA). Clin Res Cardiol. 2020 Nov;109(11):1319-1332. doi: 10.1007/s00392-020-01650-9. Epub 2020 Apr 18. PMID 32306083
- [Background] Boda-Heggemann J, Blanck O, Mehrhof F, Ernst F, Buergy D, Fleckenstein J, Tulumen E, Krug D, Siebert FA, Zaman A, Kluge AK, Parwani AS, Andratschke N, Mayinger MC, Ehrbar S, Saguner AM, Celik E, Baus WW, Stauber A, Vogel L, Schweikard A, Budach V, Dunst J, Boldt LH, Bonnemeier H, Rudic B. Interdisciplinary Clinical Target Volume Generation for Cardiac Radioablation: Multicenter Benchmarking for the RAdiosurgery for VENtricular TAchycardia (RAVENTA) Trial. Int J Radiat Oncol Biol Phys. 2021 Jul 1;110(3):745-756. doi: 10.1016/j.ijrobp.2021.01.028. Epub 2021 Jan 27. PMID 33508373
- [Background] Krug D, Blanck O, Andratschke N, Guckenberger M, Jumeau R, Mehrhof F, Boda-Heggemann J, Seidensaal K, Dunst J, Pruvot E, Scholz E, Saguner AM, Rudic B, Boldt LH, Bonnemeier H. Recommendations regarding cardiac stereotactic body radiotherapy for treatment refractory ventricular tachycardia. Heart Rhythm. 2021 Dec;18(12):2137-2145. doi: 10.1016/j.hrthm.2021.08.004. Epub 2021 Aug 8. PMID 34380072
- [Background] Kluge A, Ehrbar S, Grehn M, Fleckenstein J, Baus WW, Siebert FA, Schweikard A, Andratschke N, Mayinger MC, Boda-Heggemann J, Buergy D, Celik E, Krug D, Kovacs B, Saguner AM, Rudic B, Bergengruen P, Boldt LH, Stauber A, Zaman A, Bonnemeier H, Dunst J, Budach V, Blanck O, Mehrhof F. Treatment Planning for Cardiac Radioablation: Multicenter Multiplatform Benchmarking for the RAdiosurgery for VENtricular TAchycardia (RAVENTA) Trial. Int J Radiat Oncol Biol Phys. 2022 Jun 15;114(2):360-372. doi: 10.1016/j.ijrobp.2022.06.056. PMID 35716847
- [Background] Mayinger M, Boda-Heggemann J, Mehrhof F, Krug D, Hohmann S, Xie J, Ehrbar S, Kovacs B, Merten R, Grehn M, Zaman A, Fleckenstein J, Kaestner L, Buergy D, Rudic B, Kluge A, Boldt LH, Dunst J, Bonnemeier H, Saguner AM, Andratschke N, Blanck O, Schweikard A. Quality assurance process within the RAdiosurgery for VENtricular TAchycardia (RAVENTA) trial for the fusion of electroanatomical mapping and radiotherapy planning imaging data in cardiac radioablation. Phys Imaging Radiat Oncol. 2022 Dec 26;25:100406. doi: 10.1016/j.phro.2022.12.003. eCollection 2023 Jan. PMID 36655216
- [Background] Hohmann S, Xie J, Eckl M, Grehn M, Karfoul N, Janorschke C, Merten R, Rudic B, Buergy D, Lyan E, Krug D, Mehrhof F, Boldt LH, Corradini S, Fanslau H, Kaestner L, Zaman A, Giordano FA, Duncker D, Dunst J, Tilz RR, Schweikard A, Blanck O, Boda-Heggemann J. Semi-automated reproducible target transfer for cardiac radioablation - A multi-center cross-validation study within the RAVENTA trial. Radiother Oncol. 2024 Nov;200:110499. doi: 10.1016/j.radonc.2024.110499. Epub 2024 Sep 4. PMID 39242029
- [Result] Krug D, Zaman A, Eidinger L, Grehn M, Boda-Heggemann J, Rudic B, Mehrhof F, Boldt LH, Hohmann S, Merten R, Buergy D, Fleckenstein J, Kluge A, Rogge A, Both M, Rades D, Tilz RR, Olbrich D, Konig IR, Siebert FA, Schweikard A, Vonthein R, Bonnemeier H, Dunst J, Blanck O. Radiosurgery for ventricular tachycardia (RAVENTA): interim analysis of a multicenter multiplatform feasibility trial. Strahlenther Onkol. 2023 Jul;199(7):621-630. doi: 10.1007/s00066-023-02091-9. Epub 2023 Jun 7. PMID 37285038
- [Result] Kaestner L, Boda-Heggemann J, Fanslau H, Xie J, Schweikard A, Giordano FA, Blanck O, Rudic B. Electroanatomical mapping after cardiac radioablation for treatment of incessant electrical storm: a case report from the RAVENTA trial. Strahlenther Onkol. 2023 Nov;199(11):1018-1024. doi: 10.1007/s00066-023-02136-z. Epub 2023 Sep 12. PMID 37698592
- [Result] Mehrhof F, Huttemeister J, Tanacli R, Bock M, Bogner M, Schoenrath F, Falk V, Zips D, Hindricks G, Gerds-Li JH, Hohendanner F. Cardiac radiotherapy transiently alters left ventricular electrical properties and induces cardiomyocyte-specific ventricular substrate changes in heart failure. Europace. 2023 Dec 28;26(1):euae005. doi: 10.1093/europace/euae005. PMID 38193546